CLINICAL TRIAL: NCT06864117
Title: Comparison of Urine Flow Measurements in the Context of Pressure Flow Studies in Men in Supine and Sitting Positions Using a Urinary Condom
Brief Title: Urodynamics: Prone Vs. Seated Position
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kantonsspital Winterthur KSW (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2024-01522
Record Dates: First submitted 2025-02-25; First posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Urodynamic Studies; Urodynamics; Outlet Obstruction
Keywords: obstruction; urodynamics
MeSH Terms: conditions — Bites and Stings

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A: sitting, lying down(s/l) (Other)
  Interventions: Other: Body position during urodynamics
- Goup B: lying down, sitting (l/s) (Other)
  Interventions: Other: Body position during urodynamics

INTERVENTIONS:
Other: Body position during urodynamics — The group defines the body position in which the first and second measurements are taken.
  Group A: sitting, lying down (s/l). Group B: lying down, sitting (l/s). According to the ICS standard, the third measurement is always taken in a sitting position.

SUMMARY:
To demonstrate the feasibility of a pressure-flow study using a urinary condom with drainage tube in the sitting and lying position in everyday clinical practice and the comparability of the measured values with the "conventional" pressure-flow studies according to the ICS standard with regard to the diagnosis of outlet obstruction in men.

DETAILED DESCRIPTION:
The study aims to investigate a change in the measured values of a pressure-flow measurement in male patients between the sitting and lying position using a urinary condom. This offers enormous added value for science, as both a technique for carrying out the measurement and the effect of positioning can be evaluated. Due to anatomical conditions, this project will only be carried out with male patients. By carrying out the individual measurements in different examination positions on the same patient, influences caused by the change in position can be verified. It enables direct comparison of the criteria for outlet obstruction in the same patient and thus leads to confirmation or rejection of the hypothesis that the outlet obstruction criteria can be used for measurements in the supine position in the same way as for the measurement in the sitting position described by ICS. This project is therefore based on the question of whether the known analysis criteria for outlet obstruction are equivalent to the measurements recommended by ICS in the sitting position in male patients in whom pressure-flow studies can only be performed in the supine position. In addition, the use of a urinal condom with a drainage line as an aid or technique during the measurement is being investigated.

ELIGIBILITY:
Inclusion Criteria:

* Genotype and phenotype XY
* Age between 18 and 90 years
* Signed informed consent form
* Ability to understand and follow the study procedures and understand the consent form
* possibility ti carry out out the necessary urodynamics as part of the regular clinical examination
* assessment of neurogenic and/or non-neurogenic (idiopathic) bladder dysfunction
* Spontaneous micturition in a sitting position is possible

Exclusion criteria:

* Patients with assistance/patients under guardianship
* Patients with latex allergy or cross-allergy (banana, kiwi, fig, avocado)
* No spontaneous movement possible in a sitting position
* Sitting position not possible due to lack of trunk stability/circulatory problems
* Intravesical Botox injection during the last 9 months

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-02-28 (Estimated); Primary Completion 2028-02-28 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
First sensation of filling, FSF [mL] | Periprocedural
  measured during storage phase
First desire to void, FDV [mL] | Periprocedural
  measured during storage phase
Strong desire to void, SDV [mL] | Periprocedural
  measured during storage phase
Pdet(S) [cmH2O] | Periprocedural
  Maximum detrusor pressure, measured during storage phase
Electromyography pelvic floor EMG [μV] during storage phase | Periprocedural
Filling volume [mL] during storage phase | Periprocedural
Compl [mL/cmH2O] | Periprocedural
  Compliance, measured during storage phase
Maximum detrusor pressure during the voiding phase (Pdet(E) [cmH2O]) | Periprocedural
Detrusor pressure at maximum flow rate (PdetQmax [cmH2O]) | Periprocedural
  measured during voiding phase
Maximum flow rate (Qmax [mL/s]) during voiding phase | Periprocedural
Electromyography pelvic floor (EMG [μV]) during voiding phase | Periprocedural
Flow volume [mL] during voiding phase | Periprocedural
Residual urine volume (post void residual, PVR [mL]) | Periprocedural